CLINICAL TRIAL: NCT05815290
Title: A Phase II Trial of Cadonilimab in Locally Advanced Stage II/III MSI-H/dMMR Colorectal Cancer
Brief Title: Cadonilimab in Locally Advanced MSI-H/dMMR Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3626
Record Dates: First submitted 2023-04-01; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: dMMR Colorectal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dMMR/MSI-H colon cancer (Experimental)
  Interventions: Drug: Cadonilimab
- dMMR/MSI-H rectal cancer (Experimental)
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab 10mg/kg iv on day 1 for every 21 days with a total of 8 cycles

SUMMARY:
This is a two-arm phase II clinical study to evaluate the efficacy and safety of Cadonilimab (a PD-1/CTLA-4 bispecific antibody) in MSI-H/dMMR locally advanced colorectal cancer as the regimen of neoadjuvant treatment. Eligible patients will receive Cadonilimab monotherapy for eight cycles before surgery and part of patients may exempt from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1: Histologically or pathologically confirmed colon adenocarcinoma with a stage of T3-4 or N+ according to the CT or endoscope; Arm 2: Histologically or pathologically confirmed rectal adenocarcinoma located within 12cm from the anus with a stage of T2-4 or N+ according to the CT or endoscope
* Sign the informed consent form
* 18 years and older
* Mismatch repair deficient determined by immunohistochemistry or microsatellite instable by PCR
* No prior treatment
* Performance status: ECOG 0-1
* Good organ function:

Blood routine: hemoglobin ≥90g/L, neutrophil ≥1.5×10^9/L, platelet ≥80×10^9/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥50ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL; Ejection fraction at least 50% (or lower limit of normal) by echocardiogram

Exclusion Criteria:

* Other pathological category, such as squamous cancer
* Distant metastasis or peritoneum implantation
* Have received chemotherapy or radiotherapy in the past
* Known to have allergic reactions to any ingredients or excipients of experimental drugs
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment
* Have received colorectal cancer surgery
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C
* Pregnant or nursing
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results
* There are other serious diseases that the researchers believe patients cannot be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 3 years
  For colon cancer arm, complete response rate include the rate of pathological complete response and clinical complete response; for rectal cancer arm, complete response rate means the rate of clinical complete response

SECONDARY OUTCOMES:
OS | From date of initiation of treatment to date of death due to any cause, assessed up to 3 years
  Overall survival
DFS | From date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 3 years
  Disease free survival
pCR rate | 2 year
  The rate of pathologic complete response for patients receiving surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No